CLINICAL TRIAL: NCT03661333
Title: Dissemination and Implementation Field Trial of Dialectical Behavior Therapy for Adolescents With Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Dr. Benjamin Goldstein, Senior Scientist, Psychiatrist, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 042-2018
Record Dates: First submitted 2018-08-31; First posted 2018-09-07 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Bipolar Disorder
Keywords: dialectical behavior therapy
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adolescents with bipolar disorder (Experimental): 40 adolescents aged 13 to 19 with bipolar disorder (type I, type II, not otherwise specified/nos) will be enrolled in the dialectical behavioral therapy intervention.
  Interventions: Behavioral: Dialectical behavioral therapy

INTERVENTIONS:
Behavioral: Dialectical behavioral therapy — DBT will be conducted over 1 year, and divided into two modalities: skills training, conducted in 60 minute biweekly family meetings and individual therapy conducted in 60 minute biweekly sessions. Family skills training proceeds as follows: psychoeducation about DBT and bipolar disorder, mindfulness skills, emotion regulation skills, distress tolerance skills, interpersonal skills, and walking the middle path skills. Individual therapy sessions aim to aid the adolescent in applying skills in their daily lives. We adopt the standard DBT hierarchy of treatment targets, whereby the individual therapist selects behaviors to focus on based on the following priorities: 1) decreasing life-threatening behaviors, 2) decreasing therapy-interfering behaviors, 3) decreasing quality-of-life interfering behaviors, and 4) increasing behavioral skills. Therapists will be available to participants and their participating family members by cell phone for in-vivo skills coaching between sessions.
  Other Names: DBT

SUMMARY:
The overarching goal of this project is to evaluate the feasibility of implementing dialectical behavior therapy DBT for adolescents with bipolar disorder in an outpatient mental health clinic. In collaboration with the University of Pittsburgh, this study will measure study therapists' knowledge of the DBT model, adherence to the treatment model, and satisfaction with the treatment model.

DETAILED DESCRIPTION:
This study proposes to implement dialectical behavior therapy (DBT) for adolescents with bipolar disorder (BD) in an outpatient mental health clinic serving youth with bipolar spectrum disorders. In collaboration with the University of Pittsburgh, this study will systemically operationalize, implement, and examine the specific training, supervision, and programmatic systems needed to successfully implement and sustain the intervention in an adherent manner to achieve positive patient outcomes. This study therefore presents a unique opportunity to enhance understanding of the necessary procedures for implementing the treatment in the community, while allowing us to examine effectiveness of the intervention at the community level.

Aim 1: To examine the short- and longer-term feasibility and acceptability of a training program in DBT for adolescents with BD through clinician satisfaction ratings.

Aim 2: To examine the short- and longer-term effects of the training on practitioner knowledge and performance, and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Age 13 years, 0 months to 19 years, 11 months
* Meet diagnostic criteria for BD by KSADS-PL
* Engaged in, or willing to proceed with, a pharmacotherapy regimen
* At least one parent/guardian with whom the patient lives or regularly interacts (>5 hours per week) is willing to participate in skills training
* Able and willing to give informed consent/assent to participate.

Exclusion Criteria:

* Evidence of mental retardation, moderate to severe pervasive developmental disorder, or organic central nervous system disorder by the K-SADS-PL, parent report, medical history, or school records
* A life-threatening medical condition requiring immediate treatment
* Current victim of sexual or physical abuse.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2021-11-08 (Actual)

PRIMARY OUTCOMES:
Therapist satisfaction and acceptability | Baseline
  Therapists will complete a questionnaire (Therapist Satisfaction and Acceptability Questionnaire) assessing their satisfaction with the training and treatment approach at 6 months. Acceptability will be defined as mean acceptability ratings > 5 ("acceptable") on a likert scale from 1 ("very unacceptable") to 7 ("very acceptable").
Therapist satisfaction and acceptability | 6 months
  Therapists will complete a questionnaire (Therapist Satisfaction and Acceptability Questionnaire) assessing their satisfaction with the training and treatment approach at 6 months. Acceptability will be defined as mean acceptability ratings > 5 ("acceptable") on a likert scale from 1 ("very unacceptable") to 7 ("very acceptable").
therapists will adhere to the DBT Adherence Rating Scale | End of study year 2
  Tapes will be rated for adherence using the DBT Adherence Rating scale. The scale generates a Global Score of DBT adherence and subscale scores for the 12 DBT strategy domains. To examine sustained adherence, each therapist will submit 3 consecutive sessions for adherence coding. The rating scale is not available to the public and is utilized by the DBT-Linehan Board of Certification (copyright). Please see http://www.dbt-lbc.org/downloads/Applicant_Handbook_final_with_RW_review_2018.pdf for more information.
Therapists will obtain a passing grade of the DBT Certification Exam | 1 year
  Clinicians will attain knowledge and fidelity required to pass the DBT certification examination (exam total score ≥ 80%; passing score on case conceptualization; two of three consecutive tapes coded at or above adherence). Please see the certification manual http://www.dbt-lbc.org/downloads/Applicant_Handbook_final_with_RW_review_2018.pdf for more information.
Therapist satisfaction and acceptability | 12 months
  Therapists will complete a questionnaire (Therapist Satisfaction and Acceptability Questionnaire) assessing their satisfaction with the training and treatment approach at 12 months. Acceptability will be defined as mean acceptability ratings > 5 ("acceptable") on a likert scale from 1 ("very unacceptable") to 7 ("very acceptable").
Therapist satisfaction and acceptability | 24 months
  Therapists will complete a questionnaire (Therapist Satisfaction and Acceptability Questionnaire) assessing their satisfaction with the training and treatment approach at 24 months. Acceptability will be defined as mean acceptability ratings > 5 ("acceptable") on a likert scale from 1 ("very unacceptable") to 7 ("very acceptable").

SECONDARY OUTCOMES:
Change in symptoms using the Longitudinal Interval Follow-up Evaluation (LIFE) | Baseline to 6 months
  The Longitudinal Interval Follow-up Evaluation (LIFE) will provide a comprehensive cross-sectional and longitudinal picture of the symptomatic and psychosocial course and outcome of all participants in this study. Scores range from 0-3 on certain disorders and 0-6 for other disorders. High scores indicate high level of symptom impairment.
Change in symptoms using the Longitudinal Interval Follow-up Evaluation (LIFE) | 6 months to 12 months
  The Longitudinal Interval Follow-up Evaluation (LIFE) will provide a comprehensive cross-sectional and longitudinal picture of the symptomatic and psychosocial course and outcome of all participants in this study. Scores range from 0-3 on certain disorders and 0-6 for other disorders. High scores indicate high level of symptom impairment.
Schedule for Affective Disorders and Schizophrenia for School Age Children, Present and Life Version (K-SADS-PL) | Baseline
  The K-SADS-PL is a semi-structured interview designed to ascertain present episode and lifetime history of psychiatric illness, according to Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV criteria for children and adolescents.
K-SADS Mania Rating Scale (MRS) | Baseline
  The K-SADS MRS is a 13-item rating scale with scores ranging from 0 to 6. In addition to assessing common manic symptoms, it includes the K-SADS-PL items that assess the presence and severity of hallucinations and delusions.
Depression section of the K-SADS-Present Episode Version (K-SADS-Dep) | Baseline
  The K-SADS-Dep will be used to assess the presence and severity of depressive symptoms. It is a 21-item semi-structured interview that allows depression symptom severity to be rated on a 6-point scale, from none to severe.
Change in hypo/mania symptoms using the Child Mania Rating Scale (CMRS) | Baseline to 3 months
  Parent and adolescent reported depressive and manic symptoms will be measured via the CMRS. The CMRS is a valid 21-item screening instrument, reflecting the DSM-IV criteria for a manic episode, with each response rated on a four-point Likert-type scale.
Change in hypo/mania symptoms using the Child Mania Rating Scale (CMRS) | 3 months to 6 months
  Parent and adolescent reported depressive and manic symptoms will be measured via the CMRS. The CMRS is a valid 21-item screening instrument, reflecting the DSM-IV criteria for a manic episode, with each response rated on a four-point Likert-type scale.
Change in hypo/mania symptoms using the Child Mania Rating Scale (CMRS) | 6 months to 9 months
  Parent and adolescent reported depressive and manic symptoms will be measured via the CMRS. The CMRS is a valid 21-item screening instrument, reflecting the DSM-IV criteria for a manic episode, with each response rated on a four-point Likert-type scale.
Change in hypo/mania symptoms using the Child Mania Rating Scale (CMRS) | 9 months to 12 months
  Parent and adolescent reported depressive and manic symptoms will be measured via the CMRS. The CMRS is a valid 21-item screening instrument, reflecting the DSM-IV criteria for a manic episode, with each response rated on a four-point Likert-type scale.
Change in suicidality using the Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline to 6 months
  We will assess suicidal events (past and over follow-up) with the Pediatric Version of the C-SSRS. The C-SSRS has sound psychometric properties, yields ratings of widely accepted definitions of youth suicidal events, and was used in other pediatric treatment trials yielding standardized outcomes to compare across studies. This is a semi-structured interview that includes yes/no questions as well as narrative. It captures number of suicidal events as well as type and severity.
Change in suicidality using the Columbia-Suicide Severity Rating Scale (C-SSRS) | 6 months to 12 months
  We will assess suicidal events (past and over follow-up) with the Pediatric Version of the C-SSRS. The C-SSRS has sound psychometric properties, yields ratings of widely accepted definitions of youth suicidal events, and was used in other pediatric treatment trials yielding standardized outcomes to compare across studies. This is a semi-structured interview that includes yes/no questions as well as narrative. It captures number of suicidal events as well as type and severity.
Change in symptoms using the Mood and Feelings Questionnaire (MFQ) | Baseline to 3 months,
  Self-reported depressive and manic symptoms will be measured via the MFQ. Responses are made on a 3-point scale ("0=not true", "1=sometimes true" and "2=true").
Change in symptoms using the Mood and Feelings Questionnaire (MFQ) | 3 months to 6 months
  Self-reported depressive and manic symptoms will be measured via the MFQ. Responses are made on a 3-point scale ("0=not true", "1=sometimes true" and "2=true").
Change in symptoms using the Mood and Feelings Questionnaire (MFQ) | 6 months to 9 months
  Self-reported depressive and manic symptoms will be measured via the MFQ. Responses are made on a 3-point scale ("0=not true", "1=sometimes true" and "2=true").
Change in symptoms using the Mood and Feelings Questionnaire (MFQ) | 9 months to 12 months
  Self-reported depressive and manic symptoms will be measured via the MFQ. Responses are made on a 3-point scale ("0=not true", "1=sometimes true" and "2=true").
Change in suicidality using the Suicidal Ideation Questionnaire (SIQ) | Baseline to 3 months
  Adolescents will also complete the self-report SIQ, which is intended to identify adolescents whose level of suicidal ideation is severe enough to warrant further intervention. Each item is rated on a 7-point Likert-type scale (0= "I never had this thought" to 6="almost every day") and is used to indicate the frequency with which the adolescent experiences each thought.
Change in suicidality using the Suicidal Ideation Questionnaire (SIQ) | 3 months to 6 months
  Adolescents will also complete the self-report SIQ, which is intended to identify adolescents whose level of suicidal ideation is severe enough to warrant further intervention. Each item is rated on a 7-point Likert-type scale (0= "I never had this thought" to 6="almost every day") and is used to indicate the frequency with which the adolescent experiences each thought.
Change in suicidality using the Suicidal Ideation Questionnaire (SIQ) | 6 months to 9 months
  Adolescents will also complete the self-report SIQ, which is intended to identify adolescents whose level of suicidal ideation is severe enough to warrant further intervention. Each item is rated on a 7-point Likert-type scale (0= "I never had this thought" to 6="almost every day") and is used to indicate the frequency with which the adolescent experiences each thought.
Change in suicidality using the Suicidal Ideation Questionnaire (SIQ) | 9 months to 12 months
  Adolescents will also complete the self-report SIQ, which is intended to identify adolescents whose level of suicidal ideation is severe enough to warrant further intervention. Each item is rated on a 7-point Likert-type scale (0= "I never had this thought" to 6="almost every day") and is used to indicate the frequency with which the adolescent experiences each thought.
Change in emotion regulation using the Difficulties in Emotion Regulation Scale (DERS) | Baseline to 3 months
  Adolescents will also complete the DERS, a 36-item questionnaire assessing emotional dysregulation. Participants indicate how often each item applies to them on a scale from 1="almost never; 0-10%" to 5= "almost always; 91-100%".
Change in emotion regulation using the Difficulties in Emotion Regulation Scale (DERS) | 3 months to 6 months
  Adolescents will also complete the DERS, a 36-item questionnaire assessing emotional dysregulation. Participants indicate how often each item applies to them on a scale from 1="almost never; 0-10%" to 5= "almost always; 91-100%".
Change in emotion regulation using the Difficulties in Emotion Regulation Scale (DERS) | 6 months to 9 months
  Adolescents will also complete the DERS, a 36-item questionnaire assessing emotional dysregulation. Participants indicate how often each item applies to them on a scale from 1="almost never; 0-10%" to 5= "almost always; 91-100%".
Change in emotion regulation using the Difficulties in Emotion Regulation Scale (DERS) | 9 months to 12 months
  Adolescents will also complete the DERS, a 36-item questionnaire assessing emotional dysregulation. Participants indicate how often each item applies to them on a scale from 1="almost never; 0-10%" to 5= "almost always; 91-100%".
Treatment Satisfaction Questionnaire (18-item) | 12 months
  Following the year-long DBT intervention, patients and parents will complete an 18-item Treatment Satisfaction Questionnaire. This assesses clients' satisfaction of the service (responses range from quite dissatisfied to very satisfied) as well as whether or not the service addressed the clients' needs.
Treatment Satisfaction Questionnaire (18-item) | 3 months
  Following the year-long DBT intervention, patients and parents will complete an 18-item Treatment Satisfaction Questionnaire. This assesses clients' satisfaction of the service (responses range from quite dissatisfied to very satisfied) as well as whether or not the service addressed the clients' needs.
Treatment Satisfaction Questionnaire (18-item) | 6 months
  Following the year-long DBT intervention, patients and parents will complete an 18-item Treatment Satisfaction Questionnaire. This assesses clients' satisfaction of the service (responses range from quite dissatisfied to very satisfied) as well as whether or not the service addressed the clients' needs.
Change in symptoms using the Structured Interview for DSM-IV Personality (SIDP-IV): Borderline Personality Disorder | Baseline to 6 months
  Borderline and antisocial personality symptoms will be assessed using the Structured Interview for DSM-IV Personality. The SID-P uses a semi structured interview format to assess for symptoms of personality disorders.
Change in symptoms using the Structured Interview for DSM-IV Personality (SIDP-IV): Borderline Personality Disorder | 6 months to 12 months
  Borderline and antisocial personality symptoms will be assessed using the Structured Interview for DSM-IV Personality. The SID-P uses a semi structured interview format to assess for symptoms of personality disorders.
Change in affective lability using the Children's Affective Lability Scale (CALS) | Baseline to 3 months
  The CALS is a reliable 20-item adolescent- and parent-reported measure of mood lability, derived from the adult Affective Lability Scale that was specifically designed for adults with BD. It yields a total score as well as an angry/depressed factor and a disinhibited/impersistent factor.
Change in affective lability using the Children's Affective Lability Scale (CALS) | 3 months to 6 months
  The CALS is a reliable 20-item adolescent- and parent-reported measure of mood lability, derived from the adult Affective Lability Scale that was specifically designed for adults with BD. It yields a total score as well as an angry/depressed factor and a disinhibited/impersistent factor.
Change in affective lability using the Children's Affective Lability Scale (CALS) | 6 months to 9 months
  The CALS is a reliable 20-item adolescent- and parent-reported measure of mood lability, derived from the adult Affective Lability Scale that was specifically designed for adults with BD. It yields a total score as well as an angry/depressed factor and a disinhibited/impersistent factor.
Change in affective lability using the Children's Affective Lability Scale (CALS) | 9 months to 12 months
  The CALS is a reliable 20-item adolescent- and parent-reported measure of mood lability, derived from the adult Affective Lability Scale that was specifically designed for adults with BD. It yields a total score as well as an angry/depressed factor and a disinhibited/impersistent factor.
Dialectical Behavior Therapy Barriers to Implementation | Baseline to 6 months
  The Dialectical Behavior Therapy Barriers to Implementation (DBT-BTI) is a 26-item self-report survey that assesses barriers to DBT implementation in four domains: team, direction/motivation, theoretical position/philosophy, and administrative/structural problems. It is a yes/no questionnaire and higher scores indicate higher challenges in implementation. To be completed by DBT therapist participants.
Dialectical Behavior Therapy Barriers to Implementation | 6 months to 12 months
  The Dialectical Behavior Therapy Barriers to Implementation (DBT-BTI) is a 26-item self-report survey that assesses barriers to DBT implementation in four domains: team, direction/motivation, theoretical position/philosophy, and administrative/structural problems. It is a yes/no questionnaire and higher scores indicate higher challenges in implementation. To be completed by DBT therapist participants.
Dialectical Behavior Therapy Barriers to Implementation | 12 months to 24 months
  The Dialectical Behavior Therapy Barriers to Implementation (DBT-BTI) is a 26-item self-report survey that assesses barriers to DBT implementation in four domains: team, direction/motivation, theoretical position/philosophy, and administrative/structural problems. It is a yes/no questionnaire and higher scores indicate higher challenges in implementation. To be completed by DBT therapist participants.
Barriers and Facilitators Assessment Instrument (name of scale) | Baseline to 6 months
  Therapists will complete the Barriers and Facilitators Assessment Instrument which is a well-validated and widely used measure, and is the only measure available that is designed to assess barriers and facilitators at each of the levels proposed within one instrument. It is a 16 item Likert scale questionnaire ranging from 1 to 6 with some items being reverse scored. High scores generally indicate challenges to implementation.
Barriers and Facilitators Assessment Instrument (name of scale) | 6 months to 12 months
  Therapists will complete the Barriers and Facilitators Assessment Instrument which is a well-validated and widely used measure, and is the only measure available that is designed to assess barriers and facilitators at each of the levels proposed within one instrument. It is a 16 item Likert scale questionnaire ranging from 1 to 6 with some items being reverse scored. High scores generally indicate challenges to implementation.
Barriers and Facilitators Assessment Instrument (name of scale) | 12 months to 24 months
  Therapists will complete the Barriers and Facilitators Assessment Instrument which is a well-validated and widely used measure, and is the only measure available that is designed to assess barriers and facilitators at each of the levels proposed within one instrument. It is a 16 item Likert scale questionnaire ranging from 1 to 6 with some items being reverse scored. High scores generally indicate challenges to implementation.
Implementation Climate Scale | Baseline to 6 months
  The Implementation Climate Scale will enable the team to document relevant organizational processes the aid in implementation of this treatment and provide a context for other evidence-based treatment dissemination studies. This is a Likert scale from 0 to 4 with low scores indicating challenges with implementation.
Implementation Climate Scale | 6 months to 12 months
  The Implementation Climate Scale will enable the team to document relevant organizational processes the aid in implementation of this treatment and provide a context for other evidence-based treatment dissemination studies. This is a Likert scale from 0 to 4 with low scores indicating challenges with implementation.
Implementation Climate Scale | 12 months to 24 months
  The Implementation Climate Scale will enable the team to document relevant organizational processes the aid in implementation of this treatment and provide a context for other evidence-based treatment dissemination studies. This is a Likert scale from 0 to 4 with low scores indicating challenges with implementation.
Change in therapist self-assessment | Every month for two years through study completion, an average 24 months.
  The Dialectical Behavior Therapy (DBT) Therapist Self-Assessment will allow for DBT therapists to provide subjective appraisals of their own level of comfort and confidence in applying the treatment. It also assesses the need for additional supervision from the study supervisor, consultant, and/or peer. Scores range from 1 to 7 on a Likert scale and high scores indicate high therapist level of comfort in implementing the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin I Goldstein, MD, PhD, Principal Investigator — Sunnybrook Research Insitute
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No